CLINICAL TRIAL: NCT00067431
Title: A Study of the Safety and Efficacy of Depakote Sprinkle Capsules in the Treatment of Partial Seizures in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-552
Record Dates: First submitted 2003-08-19; First posted 2003-08-20 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Partial Seizure Disorder
Keywords: Partial Seizures
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Valproic Acid

INTERVENTIONS:
Drug: Divalproex Sodium (Depakote® Sprinkle Capsules)

SUMMARY:
The purpose of this study is to compare the safety and efficacy of two concentration ranges of valproate using Depakote Sprinkle Capsules as adjunctive therapy in the treatment of partial seizures, with or without secondary generalization, in children 3-10 years.

ELIGIBILITY:
INCLUSION CRITERIA:

Subject has diagnosis of partial seizures with/without secondary generalization, supported by:

* Observed ictal events consistent with partial seizures: With/ without secondary generalization; Documented by reliable observers
* 1 of following 2: EEG at some time in past demonstrating focal abnormalities consistent with partial seizures; OR, in absence of demonstrable EEG abnormality: MRI/CT scan evidence of a focal CNS lesion consistent with partial seizures
* On stable dose of 1 or 2 antiepileptic drug(s) (AED) other than valproate, for at least 1 month
* Not taking valproate or is currently receiving valproate resulting in a trough concentration of less than 40 mcg/mL
* History of at least 4 partial seizures/month in 2 months prior to screening
* Parent/caregiver is able to keep an accurate seizure diary

EXCLUSION CRITERIA:

* History of any of following: Lennox-Gastaut syndrome; Primary generalized seizures; Infantile spasms; Mixed seizure disorders including atypical absence; Myoclonic or atonic seizures; Pseudoseizures or Epilepsia Partialis Continuans (EPC)
* Has had status epilepticus in the past 6 months
* Has significant history of any of following that would confound study results: Cardiac (including clinically important abnormality on ECG); Renal; Psychiatric (including psychosurgery); Oncologic; Endocrine; Metabolic; Pancreatic; Hepatic disease (including clinical/serological history of hepatitis); Urea cycle disorder
* Has: Expanding CNS neoplasm; Active CNS infection; Demyelinating disease; Degenerative neurological disease; Progressive encephalopathy; or any Progressive CNS disease
* Has platelet count less than or equal to 100,000/mcL
* Has blood chemistry ALT/AST value(s) greater than or equal to 2 times upper limit of normal at screening
* Requires anticoagulant drug therapy
* Not expected to be able to maintain same dose of all pre-study AEDs, excluding valproate, throughout study
* Receiving systemic chemotherapy
* Has taken lamotrigine, felbamate, or pemoline, within past 3 months prior to screening
* Has been on ketogenic diet within 30 days prior to screening
* Considered by investigator to be non-responder to valproate for treatment of epilepsy (e.g., Despite adequate trial with serum concentrations of 60 mcg/mL or greater, subject continues to have inadequate seizure control)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2003-07

PRIMARY OUTCOMES:
Change from baseline in the 4-week partial seizure rate

SECONDARY OUTCOMES:
Adverse events
Laboratory data
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, M.D., Ph.D., Study Director — Medical Director
Locations (7):
- United States (7):
  - Pediatric Epilepsy & Neurology Specialist, Tampa, Florida
  - Rainbow Babies Children's Hospital, Cleveland, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - PCTI / Children's Hospital, Columbus, Ohio
  - Primary Physician's Research, Pittsburgh, Pennsylvania
  - Texas Association of Pediatric Neurology, PA, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia